CLINICAL TRIAL: NCT04923282
Title: A Double Blind, Randomized, Single Center, Single and Multiple Dose, Pharmacokinetic, Safety and Tolerability Study of Recombinant Human Alkaline Phosphatase (recAP) Administered Intravenously in Healthy Japanese Subjects
Brief Title: Recombinant Human Alkaline Phosphatase in Healthy Japanese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AM-Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AP-recAP-AKI-01-02
Record Dates: First submitted 2021-05-25; First posted 2021-06-11 (Actual); Last update posted 2022-03-14 (Actual); Status verified 2022-03

CONDITIONS: Healthy
MeSH Terms: interventions — Single Person

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1: single 1-hour IV infusion of 0.8 mg/kg recAP or placebo (Active Comparator): single 1-hour IV infusion of 0.8 mg/kg recAP or placebo
  Interventions: Biological: single 1-hour IV infusion of 0.8 mg/kg recAP; Biological: Placebo
- Group 2: single 1-hour IV infusion of 1.6 mg/kg recAP or placebo (Active Comparator): single 1-hour IV infusion of 1.6 mg/kg recAP or placebo
  Interventions: Biological: single 1-hour IV infusion of 1.6 mg/kg recAP; Biological: Placebo
- Group 3: single 1-hour IV infusion of 3.2 mg/kg recAP or placebo (Active Comparator): single 1-hour IV infusion of 3.2 mg/kg recAP or placebo
  Interventions: Biological: single 1-hour IV infusion of 3.2 mg/kg recAP; Biological: Placebo
- Group 4: 1-hour infusions of 1.6 mg/kg recAP or placebo on Days 1, 2 and 3 (Active Comparator): 1-hour infusions of 1.6 mg/kg recAP or placebo on Days 1, 2 and 3
  Interventions: Biological: 1-hour infusions of 1.6 mg/kg recAP on Days 1, 2 and 3; Biological: Placebo

INTERVENTIONS:
Biological: single 1-hour IV infusion of 0.8 mg/kg recAP — Intravenous infusion
  Arms: Group 1: single 1-hour IV infusion of 0.8 mg/kg recAP or placebo
Biological: single 1-hour IV infusion of 1.6 mg/kg recAP — Intravenous infusion
  Arms: Group 2: single 1-hour IV infusion of 1.6 mg/kg recAP or placebo
Biological: single 1-hour IV infusion of 3.2 mg/kg recAP — Intravenous infusion
  Arms: Group 3: single 1-hour IV infusion of 3.2 mg/kg recAP or placebo
Biological: 1-hour infusions of 1.6 mg/kg recAP on Days 1, 2 and 3 — Intravenous infusion
  Arms: Group 4: 1-hour infusions of 1.6 mg/kg recAP or placebo on Days 1, 2 and 3
Biological: Placebo — Intravenous infusion

SUMMARY:
Clinical Phase 1 study to investigate the pharmacokinetics and to assess the safety and tolerability of recAP after single and multiple intravenous doses in healthy Japanese subjects.

DETAILED DESCRIPTION:
This study is a randomized, double blind, parallel group, single-center trial, consisting of a single dose part and a multiple dose part in 32 healthy Japanese subjects. Since all these doses have been studied before and safety extensively evaluated in non-Japanese subjects and no ethnic sensitivity is expected, the groups can be dosed in parallel.

Part A will have 3 parallel groups of 8 male subjects with N=6 on active and N=2 on placebo per group. Following baseline assessments, a single dose of recAP will be administered by a one-hour infusion followed by samplings for pharmacokinetic evaluation and routine safety assessments.

Part B will have a single group of 8 male subjects with N=6 on active and N=2 on placebo. Following baseline assessments, recAP will be dosed on Days 1, 2 and 3 by one-hour infusions followed by samplings for pharmacokinetic evaluation and routine safety assessments.

ELIGIBILITY:
Inclusion Criteria:

1. Gender : male
2. Age : 20-55 years, inclusive
3. Body mass index (BMI) : 18.0-30.0 kg/m2, inclusive
4. Subjects must be Japanese by birth, have resided outside Japan <10 years, have parents and maternal and paternal grandparents who are Japanese, and primarily consume a Japanese diet.
5. Resting supine blood pressure at screening showing no clinically relevant deviations from normal as judged by the Principal Investigator.
6. Computerized (12-lead) ECG recording without signs of clinically relevant pathology or showing no clinically relevant deviations.
7. All values for hematology and for clinical chemistry tests of blood and urine within the normal range or showing no clinically relevant deviations as judged by the Investigator.
8. Ability and willingness to abstain from alcohol and tobacco products from 48 h prior to entry in the clinical research center until discharge.
9. Easily accessible veins for venipuncture and catheter placing.
10. Willingness to sign the written informed consent form (ICF).
11. Subjects must agree to use adequate contraception when sexually active. This applies for the time period between end of first administration and 14 days after the last administration of study drug.

Exclusion Criteria:

1. Evidence of clinically relevant pathology.
2. History of relevant drug and/or food allergies.
3. Subject has a history of clinically significant abnormalities or of any illness that, in the opinion of the study investigator, might confound the results of the study or poses an additional risk to the subject by their participation in the study.
4. Use of medication, except for acetaminophen (paracetamol), which is allowed up to 3 days before entry into the clinical research center (after that time the use of a limited amount of acetaminophen is permitted after consultation with the Principal Investigator).
5. Subject is mentally or legally incapacitated, has significant emotional problems at the time of screening visit or expected during the conduct of the study or has a history of a clinically significant psychiatric disorder over the last year.
6. Participation in a drug study within 60 days prior to drug administration.
7. Donation of more than 500 mL of blood within 60 days prior to drug administration. Donation of more than 1.5 liters of blood (for men) in the 10 months preceding the start of this study
8. Smoking more than 5 cigarettes, 1 cigar or 1 pipe daily.
9. History of alcohol abuse or drug addiction (including soft drugs like cannabis products).
10. Positive drug screen (opiates, methadone, cocaine, amphetamines, cannabinoids, barbiturates, benzodiazepines, tricyclic antidepressants) and/or alcohol breath test at Screening and/or Pre-Dose.
11. Intake of more than 14 units of alcohol per week (one unit of alcohol equals approximately 250 mL of beer, 100 mL of wine/Japanese Sake or 35 mL of spirits).
12. Positive screen on hepatitis B surface antigen (HBsAg), anti-hepatitis C virus (anti-HCV) or anti-human immunodeficiency virus (anti-HIV)-1 or anti-HIV-2 or HIV-1/2 antigen.
13. Illness within 5 days prior to (the first) drug administration.

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 34 (Actual)
Dates: Start 2021-05-07 (Actual); Primary Completion 2021-07-08 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Maximum observed recAP plasma concentration (Cmax) after single dose | Single dose 9 days treatment phase
  Blood collection for cmax evaluation daily from Day 1 to Day 9
Time to attain maximum recAP serum concentration (Tmax) after single dose | Single dose 9 days treatment phase
  Blood collection for Tmax evaluation daily from Day 1 to Day 9
Area under the plasma concentration versus time curve (AUC) after single dose | Single dose 9 days treatment phase
  Blood collection for AUC evaluation daily from Day 1 to Day 9
recAP elimination half-life ( t1/2) after single dose | Single dose 9 days treatment phase
  Blood collection for t1/2 evaluation daily from Day 1 to Day 9
Maximum observed recAP plasma concentration (Cmax) after multiple doses | Multiple doses 13 days treatment phase
  Blood collection for cmax evaluation daily from Day 1 to Day 13
Time to attain maximum recAP serum concentration (Tmax) after multiple doses | Multiple doses 13 days treatment phase
  Blood collection for Tmax evaluation daily from Day 1 to Day 13
Area under the plasma concentration versus time curve (AUC) after multiple doses | Multiple doses 13 days treatment phase
  Blood collection for AUC evaluation daily from Day 1 to Day 13
recAP elimination half-life ( t1/2) after multiple doses | Multiple doses 13 days treatment phase
  Blood collection for t1/2 evaluation daily from Day 1 to Day 13

SECONDARY OUTCOMES:
Adverse events (AEs) after single dose | Single dose 9 days treatment phase
  Any untoward medical occurrence in a subject enrolled into a clinical study regardless of its causal relationship to study drug.
Adverse events (AEs) after multiple doses | Multiple doses 13 days treatment phase
  Any untoward medical occurrence in a subject enrolled into a clinical study regardless of its causal relationship to study drug.

CONTACTS AND LOCATIONS:
Overall Officials: Annelies Legters, Study Director — AM-Pharma
Locations (1):
- P-One Clinic, Keikokai Medical Corporation, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No